CLINICAL TRIAL: NCT03194009
Title: Public Healthcare Systems and Diabetes Prevention Among People of Mexican Origin: The PRuDENTE Initiative of Mexico City.
Brief Title: PRuDENTE; Diabetes Prevention Via Exercise, Nutrition and Treatment
Acronym: PRuDENTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Ministry of Health, Mexico City (Unknown); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Simon Barquera, Director Nutrition and Health Research Center (CINyS), Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102/100/00/16
Record Dates: First submitted 2017-06-02; First posted 2017-06-21 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetic State
Keywords: diabetes; prevention; metformin; Mexico City
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Primary health care clinics will be allocated to one of the two arms of the intervention. A) lifestyle modification, B) Metformin and lifestyle modification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle Intervention (Active Comparator): The prediabetic individuals from the primary care centres that belong to this arm, will receive only recommendations for lifestyle modifications (physical activity and diet).
  Interventions: Behavioral: Lifestyle intervention
- Metformin (Active Comparator): The prediabetic individuals from the primary care centres that belong to this arm, will receive metformin treatment and lifestyle modifications recommendations (physical activity and diet).
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The patient will received metformin 1 tablet of 850mg every 12 hrs besides lifestyle modification recommendations
  Arms: Metformin
Behavioral: Lifestyle intervention — The patient will received recommendations to modify their diet and increase their physical activity every three months towards prevention of diabetes
  Arms: Lifestyle Intervention

SUMMARY:
The PRuDENTE study proposes to assess if metformin therapy a viable, efficient and cost-effective intervention to decrease the incidence of type 2 diabetes (DMT2) in adult subjects with obesity and pre-diabetes in Mexico City. Half of the individuals recruited will receive as intervention, metformin and lifestyle modification therapy and the other half will receive only lifestyle modification therapy.

DETAILED DESCRIPTION:
Diabetes in Mexico is considered a national emergency given its high prevalence, incidence, mortality and costs. Mexico has one of the highest prevalence of diabetes; in only 6 years (2000 to 2006) this prevalence increased from 7.5% to 14.4%. In 2015, 151 deaths per 100,000 inhabitants occurred in Mexico due to diabetes complications.

Metformin is a hypoglycemia drug and it´s the first line medication for the treatment of type 2 diabetes.There is currently a significant amount of evidence that metformin administration reduces the progression from pre-diabetes to diabetes and, despite its monotherapy being less effective than lifestyle changes, the good biosafety profile and low cost have made it the drug of choice in a joint treatment.

The PRuDENTE study proposes to perform this intervention in a real environment in the clinics of the first level of care of the Ministry of Health of the Government of Mexico City, in order to provide evidence about the cost-effectiveness of metformin as a public health intervention for the prevention of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Having received primary care in the chosen health center (ideally two or more visits to that clinic in the prior year).
* Subscribers to "Seguro Popular" ( Mexican national health insurance)
* Body mass index >=30 kg / m2
* Results of fasting serum glucose with values for pre-diabetes diagnosis (glucose between 100 and 125 mg / dl)

Optional:

* Family history of DMT2 (1st grade relative).
* Previous diagnosis of hypertension or dyslipidaemia.
* Have received antihypertensive medication and / or for cholesterol / lipids.
* History of gestational diabetes mellitus.

Exclusion Criteria:

* Renal insufficiency (Glomerular Filtration Rate (GFR) <30 ml/min).
* Known hepatic impairment or altered liver enzymes (aspartate aminotransferase (AST) AST or alanine aminotransferase (ALT) three times above normal values)
* Active alcoholism or drug addiction
* Allergies or previous known intolerance to exercise or metformin.
* Current pregnancy.
* Plans to leave the area in the next three years.
* Previous diagnosis of type 2 diabetes mellitus

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3060 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes. measured by HbA1c and Fasting blood glucose (FBG) | 3 years
  We define type 2 diabetes (T2D) as either FBG 100-125 mg/dl or HbA1c of >= 6.5%
Lifestyle modifications by decreasing adiposity indicators | Will be evaluated every 3 months during the 36 month period
  We will evaluate this by : weight in Kg, height in mts. They also be combined to report BMI/m2, and waist circumference
Caloric intake | Every 3 months during the 36 month period
  From food-frequency questionnaires.
Physical Activity | Every 3 months during the 36 month period
  Expresses ad the average metabolic equivalents (METs)-hours/week

SECONDARY OUTCOMES:
Implementation process outcomes at the clinic level. Using a questionnaire | 5 years
  Assess the implementation process outcomes at the clinic-, clinician- and patient-levels that will explain the observed effectiveness, and enable future efforts to adapt and disseminate the intervention model across other primary care settings. A questionnaire will be develop to assess the feasibility and limitations for the longterm implementation of this intervention
Implementation process outcomes at the clinician level. Using a questionnaire | 5 years
  A questionnaire will be develop to assess the limitations of recruitment at the clinic . As well as to evaluate the feasibility of continuing this intervention in outside patients.
Implementation process outcomes patient level. Assess via questionnaire | 5 years
  Assess the implementation process at the patient-levels using a questionnaire that show data regarding adherence to treatment and lifestyle modifications.
Cost-utility of Metformin. Measured using cost per QALYS | 5 years
  Analyse the cost-utility of the implementation of this intervention in primary-care health. Using direct and indirect health-care cost data.

CONTACTS AND LOCATIONS:
Overall Officials: Simón Barquera, MD, PhD, Principal Investigator — Instituto Nacional de Salud Pública
Locations (1):
- Centros de Salud. Secretaría de Salud Ciudad de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez LA, Barquera S, Aguilar-Salinas CA, Sepulveda-Amor J, Sanchez-Romero LM, Denova-Gutierrez E, Balderas N, Moreno-Loaeza L, Handley MA, Basu S, Lopez-Arellano O, Gallardo-Hernandez A, Schillinger D. Design of a cluster-randomized trial of the effectiveness and cost-effectiveness of metformin on prevention of type 2 diabetes among prediabetic Mexican adults (the PRuDENTE initiative of Mexico City). Contemp Clin Trials. 2020 Aug;95:106067. doi: 10.1016/j.cct.2020.106067. Epub 2020 Jun 21. PMID 32580032